CLINICAL TRIAL: NCT03782428
Title: Probiotic Effects On Clinical and Circulating Inflammatory Cytokines Status In Patients With Colorectal Cancer: A Randomised Double Blind Clinical Trial
Brief Title: An Evaluation of Probiotic in the Clinical Course of Patients With Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dr. Liyana Zaharuddin (Other)
Responsible Party: Sponsor-Investigator, Dr. Liyana Zaharuddin, Research Assistant Physiology Department, Faculty of Medicine, National University of Malaysia
Organization: National University of Malaysia (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: FPR.4/244/TRGS/2/2014/UKM/02/3; TRGS/2/2014/UKM/02/3 (Other Grant/Funding Number: Ministry of Education, Malaysia)
Record Dates: First submitted 2018-12-16; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized double-blind placebo controlled trial was performed in patients who were diagnosed with colorectal cancer and planned for colorectal resection. Four weeks postoperative, patients were randomized to receive either placebo or 3g X 1010 probiotic containing six viable microorganism of Lactobacillus and Bifidobacterium strains for six months.
Who Masked: Participant, Investigator
Masking Description: both probiotic and placebo product were labelled as either A or B and was given to the patients through simple randomization.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic group (Active Comparator): 27 participants received probiotics twice daily for six months
  Interventions: Dietary Supplement: Probiotic
- Placebo group (Placebo Comparator): 25 participants received placebo twice daily for six months
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — 30 billions colony-forming unit (CFU) of a mixture of six viable strains including 107 mg of Lactobacillus acidophilus BCMC® 12130, Lactobacillus lactis BCMC® 12451, Lactobacillus casei subsp BCMC® 12313, Bifidobacterium longum BCMC® 02120, Bifidobacterium bifidum BCMC® 02290 and Bifidobacterium infantis BCMC® 02129
  Other Names: HEXBIO
  Arms: Probiotic group
Other: Placebo — Placebo samples produced were identical to the probiotics in term of taste and texture without live microorganisms.
  Arms: Placebo group

SUMMARY:
Colorectal cancer (CRC) is the most common cancer for men and the second most common for women. Several studies have shown that gut microbiome may play a role in triggering intestinal inflammation that leads to the development of CRC. Gut microbiome is the collection of microorganisms that inhabit the gut. Therefore, manipulation of the gut microbiome via administration of probiotics may potentially improve the health and nutritional status in patients with CRC. The aims of this study are to investigate the role of probiotic functional foods in reducing CRC-related inflammatory markers and symptom alleviation.Participants will be needed to complete an information details form which includes information on age, medical history, background details and diet. Participants are required to consume the investigational product twice daily for six months. Blood samples will be collected prior to surgery and at 6th months post product consumption. These blood samples will be processed and analysed.

DETAILED DESCRIPTION:
BACKGROUND: The study aimed to determine effects of probiotic consumption containing six viable microorganisms of 3g x 1010 Lactobacillus and Bifidobacteria strains for six months on clinical outcomes and eight colorectal cancer related inflammatory cytokines level in patients with colorectal cancer. Among cytokines investigated were Tumour Necrosis Factor alpha (TNF- α), Interferon gamma (IFN-γ), Interleukin 6 (IL-6), Interleukin 10 (IL-10), Interleukin 12 (IL-12), Interleukin 17A (IL-17A), Interleukin 17-C (IL-17C) and Interleukin 22 (IL-22)

METHODS:

A randomized, double-blind, placebo controlled trial were performed involving patients who were diagnosed with colorectal cancer and planned for colorectal resection in Universiti Kebangsaan Malaysia Medical Centre (UKMMC)

SAMPLE CALCULATION:

The effect of the intervention was described using relative risks and 95% confidence intervals and per-protocol analyses will be performed. Prior data indicate that the failure rate among controls is 0.8. If the true failure rate for experimental subjects is 0.4, the study required 22 experimental subjects and 22 control subjects to be able to reject the null hypothesis that the failure rates for experimental and control subjects are equal with probability (power) 0.8. The Type I error probability associated with this test of this null hypothesis is 0.05.An uncorrected chi-squared statistic will be applied to evaluate this null hypothesis. Assuming the dropout rate of 30%, the total patients required for this interventional study for the CRC patients is 60 (30 patients for each arm).

PATIENTS CLINICAL ASSESSMENT:

Patient clinical characteristics including age, gender, smoking habits, comorbidities, cancer stage, tumour pathological subtype and site were identified. Recruited patients were randomized through simple randomization into either treated with probiotic or placebo. Trial unblinding was done upon completion of data analysis. Patients who underwent chemotherapy during the six months intervention period were reviewed and chemotherapy induced diarrhoea were evaluated based on Common Terminology Criteria for Adverse Events version 3.0 (CTCAEv3.0).

TREATMENT PRODUCT AND PROCEDURE:

Probiotics product involved in the study was HEXBIO® manufactured by B-Crobes Laboratories Sdn. Bhd., Malaysia. HEXBIO® contains 30 billions colony-forming unit (CFU) of six viable Lactobacillus and Bifidobacteria strains including 107 mg of Lactobacillus acidophilus BCMC® 12130, Lactobacillus lactis BCMC® 12451, Lactobacillus casei subsp BCMC® 12313, Bifidobacterium longum BCMC® 02120, Bifidobacterium bifidum BCMC® 02290 and Bifidobacterium infantis BCMC® 02129. Placebo samples produced were identical to the probiotics in term of taste and texture without live microorganisms. Both samples were prepared in a form of granules placed in aluminium foil sachets and kept in room temperature. HEXBIO® was labelled as AGE 1 while placebo as AGE 2.

In order to ensure post-surgery antibiotics given will not interfere with the study results, patients were instructed to consume the product four weeks after their surgeries. Patients were required to take the products orally twice daily for six months. Good compliance were considered when patients consumed more than 70% of total products given. Anything less than this was regarded as non-compliance.

BLOOD SAMPLE COLLECTION:

Prior to surgery, five mL of blood was taken from all the recruited patients. Blood was taken into BD vacutainer and allowed to clot for 30 minutes. It was then centrifuged for 15 minutes at 1000Xg where the separated serum was stored in -80°C freezer till analyzed. The steps were repeated upon completion of the six months intervention period.

Enzyme-linked immunosorbent assay (ELISA):

Serum samples were assayed using enzyme-linked immunosorbent assay (ELISA) multiplex kit according to the manufacturer guideline (R&D System Human Magnetic Luminex Assay: LXSAHM-08).

ELIGIBILITY:
Inclusion Criteria:

* 18 years and above.
* Diagnosed with colorectal cancer
* Planned for colorectal resection

Exclusion Criteria:

* Received antibiotics 2 weeks prior to recruitment
* Consumed pro/pre/symbiotic product 2 weeks prior to recruitment,
* Patients with recurrent colorectal cancer
* Advanced metastasis
* Nursing or pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2018-11-26 (Actual)

PRIMARY OUTCOMES:
Level of circulating inflammatory cytokines (TNF-α, IFN-γ, IL-6, IL-10, IL-12, IL-17A, IL17C &IL-22) pre and post intervention. | Change from pre intervention baseline level at post six months intervention.
  the level of eight colorectal cancer related inflammatory cytokines (in pg/mL) were measured and compared between pre and post intervention in both probiotic and placebo group.

SECONDARY OUTCOMES:
Number of patients with chemotherapy induced diarrhoea assessed by CTCAE v3.0 | During the six month intervention period.
  Patients who underwent chemotherapy during the six months intervention period were reviewed and evaluated based on Common Terminology Criteria for Adverse Events version 3.0 (CTCAE v3.0).

CONTACTS AND LOCATIONS:
Overall Officials: Associate Professor Dr. Raja Affendi Raja Ali, Principal Investigator — Faculty Of Medicine, Universiti Kebangsaan Malaysia

IPD SHARING:
Plan to Share IPD: No
We are bind to the Institutional Review Board Universiti Kebangsaan Malaysia Medical Research Ethics Committee rules and regulations where recruited patients identity and data are kept confidential and will only be allowed to access by the institution.

REFERENCES:
- [Derived] Zaharuddin L, Mokhtar NM, Muhammad Nawawi KN, Raja Ali RA. A randomized double-blind placebo-controlled trial of probiotics in post-surgical colorectal cancer. BMC Gastroenterol. 2019 Jul 24;19(1):131. doi: 10.1186/s12876-019-1047-4. PMID 31340751